CLINICAL TRIAL: NCT05483153
Title: Infant-Directed Singing (IDS) for Maternal Sensitivity and Infant Self-Regulation in an At-Risk Population
Brief Title: Infant-Directed Singing for At-Risk Mothers and Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: GRAMMY Museum Grant Program (Unknown)
Responsible Party: Principal Investigator, Shannon Kay de l'Etoile, Associate Dean of Graduate Studies, Professor, Music Therapy, University of Miami
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20220297
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Maternal Behavior; Infant Behavior
MeSH Terms: conditions — Infant Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infant-Directed Singing Coaching Group (Experimental): At-risk mothers and infants will receive four, 30-minute sessions of an infant-directed singing coaching intervention.
  Interventions: Behavioral: Infant-Directed Singing Coaching

INTERVENTIONS:
Behavioral: Infant-Directed Singing Coaching — At-risk mothers will receive four, 30-minute, in-person infant-directed singing coaching intervention sessions that take place over two weeks. Mothers will learn how to better read infant cues and respond with sensitive singing. Infants will gain experience in self-regulation of arousal states.

SUMMARY:
The purpose of this study is to figure out if mothers can learn how to use singing to help their babies. Singing can help babies calm down or encourage them to play, both of which are needed for learning.

ELIGIBILITY:
Inclusion Criteria:

Mothers:

* must have infants enrolled at the Linda Ray Intervention Center (LRIC).
* must be 18 years of age or older
* must be able to read and write in English

Infants:

* must be enrolled at the Linda Ray Intervention Center (LRIC).
* must be at least 3 months and no older than 12 months.

Exclusion Criteria:

- Participants who are not enrolled at the Linda Ray Intervention Center (LRIC).

Min Age: 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-09-14 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Maternal Perceived Self-Efficacy as measured by Karitane Parenting Confidence Scale | 1 week prior to intervention, 1 week after intervention
  Change in maternal perceived self-efficacy will be measured by using the Karitane Parenting Confidence Scale. This is a 15-item self-report measure, with scores ranging from 0- 45. Lower scores reflect lower perceived self-efficacy, and higher scores indicate higher levels of perceived self-efficacy.
Change in Acoustic Parameters of Mothers' Singing | 1 week prior to intervention, week 2 of intervention, 1 week after intervention
  Change in the acoustic parameter of mothers evaluated by data mining of recording of mother's voices using a microphone
Change in percentage of time Infant displays gaze type | 1 week prior to intervention, week 2 of intervention, 1 week after intervention
  Change in percentage of time infant displays gaze type will be measured by a video recording of the infant gaze. Videos will be coded to determine the percentage of time infants demonstrate a gaze type. Types of gaze include and range from roaming (most negative), averted, neutral, intermittent, to sustained (most positive).
Change in percentage of time Infant displays affect type | 1 week prior to intervention, week 2 of intervention, 1 week after intervention
  Change in percentage of time infant displays affect type will be measured by a video recording of Infant's affect. Videos will be coded to determine the percentage of time infants demonstrate affect type. Types of affect include and range from large grimace (most negative), frown, neutral, smile, to large smile (most positive).

CONTACTS AND LOCATIONS:
Overall Officials: Shannon K de l'Etoile, PhD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Linda Ray Intervention Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No